CLINICAL TRIAL: NCT01155856
Title: Consecutive, Randomized Controlled Multicenter Trial, Investigating the Feasibility and Safety of a Telemedicine Based Treatment Regimen in Patients With Chronic Obstructive Pulmonary Disease (COPD), Compared to Conventional Hospital Treatment
Brief Title: The Virtual Hospital - a Clinical Trial
Acronym: TVH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: TRYG Foundation (Other); The TOYOTA Foundation (Unknown); Sygekassernes Helsefond (Other); Lykfeldt legat (Unknown); Frederiksberg Fonden (Unknown); Danmarks Lungeforening (Other)
Responsible Party: Principal Investigator, Klaus Phanareth, MD, ph.d, research leader, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2010-021
Record Dates: First submitted 2010-06-21; First posted 2010-07-02 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Telemedicine
Keywords: telemedicine; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemedicine (Experimental): Within 24 hours after admission for exacerbation of COPD, patients in the intervention group are sent home for further treatment (telemedicine based) instead of the conventional treatment at the hospital. Patients in the intervention group will receive the same treatment as the control group and have daily contact with the physician/nurse at the hospital through a videoconference system.
  Interventions: Other: Telemedical admission and treatment in the patients´ own homes instead of conventional admission and treatment at the hospital
- control (No Intervention): The control group will receive usual care and treatment at the hospital until discharge(typically between 5-7 days).

INTERVENTIONS:
Other: Telemedical admission and treatment in the patients´ own homes instead of conventional admission and treatment at the hospital — For this study a telemedical platform has been developed on which it is possible to treat patients in their own homes. The platform consists of a videoconference part that allows the patients to make contact to qualified medical staff and a technology part that can transfer vital indicators of the patients health condition (lung function, oxygen saturation, pulse etc.)175 patients will be included with an expected drop-out of 20 % or 35 patients. The patients will be equally recruited from two hospitals (Frederiksberg and Herlev Hospital). All patients must have an exacerbation in their COPD that requires hospitalization to be included in this study. Each patient participate in the study for 6 months after discharge with follow-up at 1, 3 and 6 months.
  Arms: telemedicine

SUMMARY:
Introduction:

With the rapid development in technology telemedicine has become a tool with the potential to improve and optimize the treatment of different diseases and to make diagnostics, treatment and counseling possible over shorter or longer distances.

Home based telemedicine is a new method that leads to a series of important questions that needs to be answered. This study is designed to answer questions concerning patient safety in telehomecare, the patients´ quality of life, efficiency and a cost benefit analysis of implementing this technology.

This study is about patients with chronic obstructive pulmonary disease (COPD) who are admitted to the hospital with an acute exacerbation. Approximately 24 hours after admission half of the patients are randomized to be admitted to their own home supported by telemedical equipment while the other half remain admitted at the hospital (typically between 5-7 days).

Primary Aim:

To investigate if telemedical surveillance and treatment in the recovery period of an acute exacerbation is just as safe as conventional admission of patients with COPD measured on treatment failure.

Secondary Aims:

To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD:

1. Is comparable in reestablishing Forced Expiratory Volume in 1 second (FEV1).
2. Demands the same number of treatment days/time before discharge/cessation of telemedical surveillance.
3. Is comparable in quality of life in the two groups of treated patients.
4. Have comparable adverse event profiles.
5. leads to a lower total cost in health services (health economical analysis)
6. Is possible to do for the patients (drop-outs because of the technical equipment or the patient does not know how to use the equipment.)

7 Is better seen from the physician's perspective when it comes to:

1. The virtual patient contact / communication
2. Technology
3. The work process compared to the conventional work process
4. Time spent with the patient
5. Usability
6. Improvement potentials ("the doctors view")

   8. The equipment is satisfactory for the patient to use

   Method

   For this study a telemedical platform has been developed on which it is possible to treat patients in their own homes. The platform consists of a videoconference part that allows the patients to make contact to qualified medical staff and a technology part that can transfer vital indicators of the patients´ health condition (lung function, oxygen saturation, pulse etc.) 175 patients will be included with an expected drop-out of 20 % or 35 patients. The patients will be equally recruited from two hospitals (Frederiksberg and Herlev Hospital). All patients must have an exacerbation in their COPD that requires hospitalization to be included in this study. Each patient participates in the study for 6 months after discharge with follow-up at 1, 3 and 6 months.

DETAILED DESCRIPTION:
In addition to the main study, two sub studies will be conducted, using the same intervention and subjects as the main study;

1. COPD patients´ self-efficacy after virtual admission compared to hospital admission - implications for clinical practice
2. Cognitive function and daily life after virtual admission compared to conventional hospital admission in patients with chronic obstructive pulmonary disease (COPD)

   --------------------------------------------------------------------------------

   Ad. 1: COPD patients´ self-efficacy after virtual admission compared to hospital admission - implications for clinical practice

   Background:

   In order to transfer the patient from the hospital to the telemedicine based homecare treatment regimen, the patient must be able to perform tests and treatments and also contribute to identification of problems and changes in the physical condition. However, so far it has not been investigated whether patients using telehomecare have or acquire the necessary skills to cope with the problems entailed by COPD, in interaction with healthcare professionals and relatives.

   Aim:

   The primary aim of this sub study is to describe what characterizes COPD patients´ self-efficacy after virtual admission compared to hospital admission.

   Method:

   Self-efficacy will be measured using "The COPD self-efficacy scale", developed by Wigal et al (Chest 1991). The mean score will be compared between the two study arms, and furthermore the changes within the two groups will be assessed. Data will be collected at baseline, and also three days, six weeks and three months after discharge.

   In addition, analyses will be conducted to explore the association between self-efficacy, readmission and the use of bed days during a three month follow-up period.

   --------------------------------------------------------------------------------

   Ad.2: Cognitive function and daily life after virtual admission compared to conventional hospital admission in patients with chronic obstructive pulmonary disease (COPD)

   Background:

   COPD affects distant organs and causes several complications, including cognitive dysfunction. The impairment forms a significant clinical problem with consequences for the patients such as dependency on help for basic daily activities, increased symptom experience and poor compliance with medical treatment.

   Aim:

   The aim of the study is to investigate cognitive function and daily life after virtual admission compared to conventional hospital admission in patients with COPD. The study is a part of a randomized multicenter trial, investigating the feasibility and safety of a telemedicine based treatment regime in COPD patients, compared to conventional hospital treatment (Telemedicine technology makes it possible to communicate with the patient using a video conference system connected to a telemedicine communication platform).

   Method:

   For this sub study, we consecutively include 150 patients from the multicenter trial. The primary outcome will be cognitive function evaluated by a neuropsychological test battery (ISPOCD), including verbal learning, memory capacity and attention, at discharge, and six weeks after discharge. The secondary outcomes is daily life evaluated by questionnaires including self-reported cognitive function, self-efficacy, activities of daily living, health related quality of life, anxiety and depression, at discharge, six weeks and three months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD stage III or IV according to GOLD guidelines
* >45 years of age
* Compliant patient (is able to see, hear and follow instructions)
* Estimated admission time > 2 days

Exclusion Criteria:

* X-score > 4 at randomization(need of NIV or respirator)
* severe overweight assessed by investigator
* serious comorbidity (malignancy,unstable heart disease, dysregulated diabetes or other disease that makes participation impossible)
* non-compliant patient (cannot follow simple instructions)
* fever (>38 degrees Celsius) at randomization point, in need of I.V. antibiotics assessed by investigator
* participation in another clinical trial within the last 30 days

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days, 3 months, 6 months
  To study essential safety parameters for the patients the numbers of deaths will be compared in the two groups using data from the Danish Death Registry.
readmission | 30 days, 3 months, 6 months
  Readmission can be considered as a treatment failure related to COPD and will thus be assessed in both groups by reviewing the hospital patient administration system.
need for additional Prednisolone, additional antibiotics , NIV or life support machine (respirator) | 30 days, 3 months, 6 months
Self-efficacy | 3 days
  Self-efficacy is measured using "The COPD self-efficacy scale". The scale has been validated in Danish, prior to its use in the current sub studies.
  The patients will be asked to fill in the questionnaire at baseline, and 3 days after discharge
Cognitive function | 3 days and six weeks after discharge
  Cognitive function evaluated by a neuropsychological test battery, International Study of Post Operative Cognitive Dysfunction (ISPOCD) including verbal learning, memory capacity and attention.

SECONDARY OUTCOMES:
FEV1 | 30 days, 3 months, 6 months
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD: Is comparable in reestablishing FEV1 (stable phase). This is however not possible to compare with patients that have just been diagnosed with COPD.
Admission days | 30 days
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD demands the same number of treatment days/time before discharge/cessation of telemedical surveillance
Healthrelated Quality of life | baseline, discharge, 4-6 weeks, 3 months, 6 months
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD is comparable in quality of life in the two groups of treated patients. Quality of life is measured via questionnaires (EQ-5D, CCQ, SGRQ)
Adverse event | 30 days
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD have comparable adverse event profiles
cost in health services | 30 days, 3 months, 6 months
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD leads to a lower total cost in health services (health economical analysis)
Telemedicine coping skills | 30 days
  To evaluate if telemedical surveillance and treatment in the recovery period of an acute exacerbation compared to conventional treatment of COPD is possible to do for the patients (drop-outs because of the technical equipment or the patient does not know how to use the equipment.)Intervention group only.
Patient satisfaction | 30 days
  To evaluate if the equipment is satisfactory for the patient to use (intervention group only). Assessed by questionnaire
Physicians/user satisfaction | 30 days
  To evaluate if telemedicine is better than hospital admission, seen from the physicians perspective, when it comes to:
  1. The virtual patient contact / communication
  2. Technology
  3. The work process compared to the conventional work process
  4. Amount of time spent with the patient
  5. Usability
  6. Improvement potentials ("the doctors view") assessed by questionnaire intervention group only
Number of bed days | 30 days
Self-reported cognitive function | 3 days, six weeks and three months after discharge
  Evaluated by a questionnaire: Subjective Cognitive Functioning (SCF)
Self-efficacy | up to 3 months
  Evaluated by the COPD Self Efficacy Scale (CSES). Will be evaluated at baseline, three days after discharge, and also six weeks and three months after discharge.
Activities of daily living | 3 days, six weeks and three months after discharge
  Evaluated by a questionnaire: Instrumental Activity of Daily Living (IADL)
Health related quality of life | 3 days, 6 weeks, 3 months after discharge
  Evaluated by a questionnaire: St George Respiratory Questionnaire (SGRQ)
Anxiety and Depression | 3 days, six weeks and three months after discharge
  Evaluated by a questionnaire: Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus V Phanareth, ass.professor, Study Director — Frederiksberg Hospital
Locations (1):
- Frederiksberg Hospital, Frederiksberg, Denmark

REFERENCES:
- [Derived] Jakobsen AS, Laursen LC, Ostergaard B, Rydahl-Hansen S, Phanareth KV. Hospital-admitted COPD patients treated at home using telemedicine technology in The Virtual Hospital Trial: methods of a randomized effectiveness trial. Trials. 2013 Sep 3;14:280. doi: 10.1186/1745-6215-14-280. PMID 24139548